CLINICAL TRIAL: NCT02969993
Title: Very Long Term VHI Voice Outcome After MTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016/394
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Laryngeal Paralysis
MeSH Terms: conditions — Vocal Cord Paralysis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Questionnaire (Experimental): Questionnaire to previously operated patients
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — evaluating the voice outcome by the fullfilment of the voice handicap index

SUMMARY:
Long term assesment of voice outcome after Montgomery Thyroplastie by performing a Survey of operated patients using the voice handicap index scale

ELIGIBILITY:
Inclusion Criteria:

* patients presenting UVFP of neurogenic origin treated by MTIS > 2 years before inclusion.
* No superior limit in terms of years.
* Age 18-80 years at the time of MTIS
* No other treatment before MTIS other than resorbing material injection laryngoplasty (maximum twice)
* No further voice treatment after MTIS except speech therapy.
* VHI or VHI-10 performed before MTIS and within the 6 months after MTIS. In case of multiple post-op VHI tests, only the earliest post-op. VHI test will be taken into account
* VHI tests validated for the utilized language

Exclusion Criteria:

* patient not able to answer VHI questionnaire personally
* Post MTIS new health condition affecting the voice tract and/ or the respiratory function.
* Post MTIS appearance of other voice/ vocal cord pathology

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-12; Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Voice handicap index | 2 years
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (2):
  - Cliniques universitaires Saint-Luc, Brussels Capital Region, Brussels Capital
  - CHU Namur -Mont-Godinne, Yvoir, Namur
- Valencia Medical School - Hospital General Universitario, Valencia, Levante, Spain